CLINICAL TRIAL: NCT01969006
Title: Effect of Ilioinguinal Blockage on Postoperative Pain After Laparoscopic Inguinal Herna Repair
Brief Title: Ilioinguinal Block in Laparoscopic Inguinal Hernia Repair
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Another study has been planned, so we did not initiate this one.
Sponsor: Randers Regional Hospital (Other)
Collaborators: Regionshospitalet Horsens (Other); Denmark (Unknown)
Responsible Party: Principal Investigator, Thorbjorn Sommer, Senior Surgeon phd, ass proffessor, Randers Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ILIOINGUINAL01
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2013-10

CONDITIONS: Post Operative Pain as Estimated by the Sue of the VAS Score
Keywords: inguinal hernia, postoperative pain, localanesthesia, nerve blockage
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection of Marcaine ½ % (Experimental): Injection of 40 ml of Marcaine ½ % 2 cm medial, 2 cm downwards from the Anterior Iliac Spine
  Interventions: Drug: Marcaine ½%
- Needle prick (Placebo Comparator): Needle prick 2 cm medial and 2 cm downwards from the Anterior Iliac spine
  Interventions: Procedure: Needle prick

INTERVENTIONS:
Drug: Marcaine ½%
  Arms: Injection of Marcaine ½ %
Procedure: Needle prick
  Arms: Needle prick

SUMMARY:
This study is undertaken to clarify whether intraoperative blockage with 40 ml of ½ % Marcaine© of the nerves in the ilio-inguinal canal may decrease postoperative pain after laparoscopic inguinal hernia repair.

Patients will be randomised to injection of Marcaine© og a needle prick per-operatively.

Pain will be estimated using the VAS score in:

1. the wound 2 the abdomen 3 the shoulder

Scoring will be performed:

1. pre-operatively
2. 1 hour postoperatively
3. at discharge from the hospital d day 1,2 and 3 post OP

e. 1 year post OP

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 year
2. Informed consent
3. a diagnosis of an inguinal hernia
4. ASA group ≤ 3
5. BMI ≤ 35

Exclusion Criteria:

1. Communication problems
2. No consent
3. Open procedure (not laparoscopic)
4. ASA-group 4
5. Use of Steroid or immunosuppressive tretament
6. Regular morphine use.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 1 year
  VAS score of pain from:
  1. wound
  2. abdomen
  3. shoulder

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Horsens Regions Hospital, Horsens
  - Randers regions Hospital, Randers